CLINICAL TRIAL: NCT04091217
Title: Atezolizumab in Combination With Bevacizumab in Patients With Unresectable Locally Advanced or Metastatic Mucosal Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML41186
Record Dates: First submitted 2019-09-13; First posted 2019-09-16 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-08

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab + Bevacizumab (Experimental)
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 1200 mg will be administered intravenously every 3 weeks.
  Other Names: Tecentriq
Drug: Bevacizumab — Bevacizumab 7.5 mg/kg will be administered intravenously every 3 weeks.
  Other Names: Avastin

SUMMARY:
This study will evaluate the efficacy and safety of atezolizumab in combination with bevacizumab in patients with unresectable locally advanced or metastatic mucosal melanoma.

DETAILED DESCRIPTION:
The study is divided into 2 stages. Stage I of the study is completed when 22 patients with measurable disease have been enrolled and completed ORR evaluation. If the number of responders in Stage I is more than 3, another 16 patients may be enrolled to Stage II.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed unresectable locally advanced(stage III) or metastatic(Stage IV) mucosal melanoma
* May have received prior systemic treatment or treatment naive at enrollment
* Measurable disease per RECIST v1.1
* ECOG Performance Status of 0-1
* Life expectancy >= 12 weeks
* Adequate hematologic and end-organ function
* Negative HIV test at screening
* Negative hepatitis B surface antigen test at screening
* Negative hepatitis B core antibody at screening, or positive total HBcAb test followed by quantitative hepatitis B virus DNA<500 IU/mL at screening.
* Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, and agreement to refrain from donating eggs
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm

Exclusion Criteria:

* Symptomatic or actively progressing central nervous system (CNS) metastases
* History of leptomeningeal disease
* Uncontrolled tumor-related pain
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures
* Uncontrolled or symptomatic hypercalcemia
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions: 1) Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study. 2) Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study. 3) Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only are eligible for the study provided all of following conditions are met: (i) Rash must cover < 10% of body surface area (ii) Disease is well controlled at baseline and requires only low-potency topical corticosteroids (iii) No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* Active tuberculosis
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
* History of malignancy other than melanoma within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death, such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer
* Prior allogeneic stem cell or solid organ transplantation
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
* Current treatment with anti-viral therapy for HBV
* Current, recent (within 28 days prior to initiation of study treatment) or planned treatment with any other investigational agent or participation in another clinical study with anti-cancer therapeutic intent
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months after the final dose of atezolizumab, 6 months after the final dose of bevacizumab

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- China (3):
  - Beijing Cancer Center; Renal Cancer And Melanoma Department., Beijing
  - Fujian Provincial Cancer Hospital, Fuzhou
  - Zhejiang Cancer Hospital, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Mao L, Fang M, Chen Y, Wei X, Cao J, Lin J, Zhang P, Chen L, Cao X, Chen Y, Guo J, Si L. Atezolizumab plus Bevacizumab in Patients with Unresectable or Metastatic Mucosal Melanoma: A Multicenter, Open-Label, Single-Arm Phase II Study. Clin Cancer Res. 2022 Nov 1;28(21):4642-4648. doi: 10.1158/1078-0432.CCR-22-1528. PMID 36044526

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 3 centers in China.
Pre-assignment Details: There were 20 participants who died during the follow-up period who were recorded as study completed as per the protocol.
Groups:
- Atezolizumab + Bevacizumab: Participants received 1200 mg atezolizumab by intravenous infusion every 3 weeks and/or 7.5 mg/kg bevacizumab by intravenous infusion every 3 weeks until unacceptable toxicity or loss of clinical benefit as determined by the investigator. Participants who transiently withheld or permanently discontinued either atezolizumab or bevacizumab may continue on single-agent therapy as long as the participants were experiencing clinical benefit in the opinion of the investigator.
Period: Overall Study
Arm/Group | Atezolizumab + Bevacizumab
Started (Intention-to-treat Population, all enrolled) | 43
Stage I Analysis Population | 22
Stage II Analysis Population | 38
Completed | 41
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Intention-to-treat population is defined as all enrolled participants regardless of whether they receive any assigned study drug.
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 43
Age, Continuous [Median (Full Range); unit: Years] | 61.0 [33 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 43
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the date of first treatment to the first occurrence of disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1.
Time Frame: Up to approximately 32 months
Population: Full Analysis Set (FAS) is defined as all enrolled participants who receive any amount of study treatment and evaluable for efficacy endpoints.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 40
Months | 8.21 [4.07 to 9.59]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from the date of first treatment to death from any cause.
Time Frame: Up to approximately 32 months
Population: Full Analysis Set (FAS) was defined as all enrolled participants who receive any amount of study treatment and evaluable for efficacy endpoints.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 40
Months | 24.77 [14.88 to NA] — The upper limit of the 95% confidence interval could not be estimated because there was an insufficient number of participants with events.

3. Secondary Outcome: Duration of Objective Response (DOR)
Description: DOR was defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first), as determined by the investigator according to RECIST v1.1
Time Frame: Up to approximately 32 months
Population: Only responders (CR/PR) assessed by investigator were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 18
Months | 12.42 [5.59 to 14.03]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the sum of a complete or partial response or stable disease rates as determined by the investigator according to RECIST v1.1.
Time Frame: Up to approximately 32 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 40
Percentage of Participants | 65.0 [48.32 to 79.37]

5. Secondary Outcome: Percentage of Participants With Adverse Events
Description: The percentage of participants who experienced an Adverse Event (AE) or Serious Adverse Event (SAE). Incidence, nature, and severity of Adverse Events (AE), are reported per the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v5.0).
Time Frame: From the first study drug to the data cutoff date: 31 August 2022 (up to approximately 32 months)
Population: Safety analysis set is defined as all enrolled participants who receive any amount of least one dose of any study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 43
Percentage of participants
  Percentage of participants with at least 1 AE | 95.3
  Percentage of participants with at least one Grade 3-5 AE | 25.6
  Percentage of participants with at least one AE by worst grade - Grade 1 | 41.9
  Percentage of participants with at least one AE by worst grade - Grade 2 | 27.9
  Percentage of participants with at least one AE by worst grade - Grade 3 | 23.3
  Percentage of participants with at least one AE by worst grade - Grade 4 | 0
  Percentage of participants with at least one AE by worst grade - Grade 5 | 2.3
  Percentage with at least one SAE | 20.9

6. Primary Outcome: Objective Response Rate (ORR) in the Full Analysis Set Analysis Population
Description: ORR was defined as the percentage of participants with a complete response (CR) defined as disappearance of all target lesions, or partial response (PR) defined as at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR, on two consecutive occasions >= 4 weeks apart, as determined by the investigator according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1).
Time Frame: Up to approximately 32 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Atezolizumab + Bevacizumab
Number analyzed (Participants) | 40
Percentage of participants | 45.0 [29.26 to 61.51]

ADVERSE EVENTS:
Time Frame: From the first study drug to the data cutoff date: 31 August 2022 (up to approximately 32 months)
Description: All-cause mortality reported for deaths that occurred during study based on ITT, which included all participants. Serious & other adverse events reported based on safety population, which included participants who received any amount of any component of study treatment.
Arm/Group | Atezolizumab + Bevacizumab
All-Cause Mortality (participants affected / at risk) | 20/43
Serious Adverse Events (participants affected / at risk) | 9/43
Other Adverse Events (participants affected / at risk) | 34/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Atezolizumab + Bevacizumab (N=43)
Immune-mediated hepatitis (Hepatobiliary disorders) | 2
Drug-induced liver injury (Hepatobiliary disorders) | 1
Abdominal infection (Infections and infestations) | 1
Hypophysitis (Endocrine disorders) | 2
Appendicitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Orbital infection (Infections and infestations) | 1
Epilepsy (Nervous system disorders) | 1
Post herpetic neuralgia (Nervous system disorders) | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Autoimmune lung disease (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atezolizumab + Bevacizumab (N=43)
Blood lactate dehydrogenase increased (Investigations) | 16
Blood cholesterol increased (Investigations) | 11
Aspartate aminotransferase increased (Investigations) | 10
Alanine aminotransferase increased (Investigations) | 9
Blood triglycerides increased (Investigations) | 9
Blood bilirubin increased (Investigations) | 8
Blood creatine phosphokinase increased (Investigations) | 7
Blood uric acid increased (Investigations) | 7
Gamma-glutamyltransferase increased (Investigations) | 6
Blood glucose increased (Investigations) | 5
White blood cell count decreased (Investigations) | 5
Bilirubin conjugated increased (Investigations) | 4
Weight decreased (Investigations) | 4
Blood bilirubin unconjugated increased (Investigations) | 3
Blood urea increased (Investigations) | 3
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 3
Protein urine present (Investigations) | 3
Pyrexia (General disorders) | 9 — General disorders and administration site conditions
Fatigue (General disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 5
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3
Constipation (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 6
Hypothyroidism (Endocrine disorders) | 8
Hyperthyroidism (Endocrine disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3
Hypertension (Vascular disorders) | 5
Anaemia (Blood and lymphatic system disorders) | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-07-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT04091217/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/17/NCT04091217/SAP_001.pdf